CLINICAL TRIAL: NCT02423876
Title: UW14030: Epidural Anesthesia as Part of an Enhanced Recovery Pathway in Gynecologic Surgery
Brief Title: Epidural Anesthesia Within an Enhanced Recovery Pathway in Reducing Pain in Patients Undergoing Gynecologic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW14030; NCI-2015-00395 (Registry Identifier: NCI Trial ID); 2014-1458 (Other: HS-IRB); A532820 (Other: UW Madison); SMPH\OBSTET & GYNEC\GYNEC ONC (Other: UW Madison); Protocol Version 11/14/2016 (Other: UW Madison)
Record Dates: First submitted 2015-04-14; First posted 2015-04-22 (Estimated); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Intraoperative Complication; Malignant Female Reproductive System Neoplasm; Pain
MeSH Terms: conditions — Intraoperative Complications; Pain | interventions — Analgesia, Epidural; Anesthesia, Epidural; Hydromorphone; Ropivacaine; Analgesia; Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (epidural placement, ERP) (Experimental): Patients undergo epidural placement in the First Day Surgery pre-operative area or similar areas suitable for insertion of epidural catheters. In the post-operative anesthesia care unit, patients may receive medication via the epidural on an as needed basis, as determined by the anesthesia team. Dosing and rate of standardized medication will be managed by the anesthesia team until the epidural is removed. Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.
  Interventions: Drug: Epidural analgesia; Other: Intraoperative Complication Management and Prevention; Procedure: Pain Therapy
- Arm II (ERP) (Active Comparator): Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.
  Interventions: Other: Intraoperative Complication Management and Prevention; Procedure: Pain Therapy

INTERVENTIONS:
Drug: Epidural analgesia — Receive epidural placement. Standard epidural medications and dosage are as follows:
  * 0.1% ropivicaine + 10 mcg/mL hydromorphone at 6 mL/hr continuous rate
  * 3 mL/hr RN bolus, to be used as needed based on pain ratings
  * 3 mL/30 minutes patient bolus, which is available on patient demand.
  Other Names: Epidural Block; ropivicaine; hydromorphone; Naropin; Dilaudid; Exalgo
  Arms: Arm I (epidural placement, ERP)
Other: Intraoperative Complication Management and Prevention — Undergo ERP
  Other Names: Intraoperative Complication Management/Prevention
Procedure: Pain Therapy — Undergo ERP
  Other Names: Analgesia; Pain Control; Pain Management; Pain, Pain Management

SUMMARY:
This randomized clinical trial studies epidural anesthesia within an enhanced recovery pathway (ERP) in reducing pain in patients undergoing gynecologic surgery. An epidural analgesia (pain relief) is a small tube placed in the lower back that numbs the nerves and stops the feeling of pain. It stays in place for several days after surgery and may be helpful for pain control in patients with gynecologic cancer after surgery. ERP is a set of specific steps used before, during, and after surgery by health care providers to care for patients after surgery. ERPs include patient education, not using laxatives before surgery, increasing activity after surgery, and scheduled use of medications for pain and nausea. Giving epidural anesthesia as part of an ERP may improve pain control in patients undergoing gynecologic surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Mean postoperative pain score for the first 24 hours post-operatively, (measured by the Numeric Rating Scale [NRS], which rates pain on a 1-10 scale, collected routinely on the post-operative floor) will be compared between the epidural and no-epidural groups.

SECONDARY OBJECTIVES:

I. Total opioid use measured in oral morphine equivalents for the first two days post-surgery.

II. Length of hospital stay (measured in hours from admission to time of discharge order placement).

III. Post-operative antiemetic use and number of recorded episodes of emesis. IV. Return of bowel function (measured in hours from completion of surgery to passage of flatus).

V. Subject satisfaction at the 4 week post-operative visit (as measured by two pain satisfaction questions taken from the Hospital Consumer Assessment of Healthcare Providers and Systems [HCAHPS] survey).

VI. Post-operative complications (urinary tract infections [UTIs], thromboembolic events, pneumonia, blood transfusion, myocardial infarction, falls).

VII. Readmission rate. VIII. Epidural discontinuation rates prior to planned removal (in epidural group only).

IX. Stress and inflammation serum and saliva markers at baseline and the first day after surgery, as well as at their postoperative visit.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo epidural placement in the First Day Surgery pre-operative area or similar areas suitable for insertion of epidural catheters. In the post-operative anesthesia care unit, patients may receive medication via the epidural on an as needed basis, as determined by the anesthesia team. Dosing and rate of standardized medication will be managed by the anesthesia team until the epidural is removed. Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.

ARM II: Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gynecologic surgery via midline vertical laparotomy at University of Wisconsin Hospital and Clinics (UWHC)
* Patients must be English speaking
* Patients must have the ability to understand visual and verbal pain scales
* Patients must be eligible for epidural placement

Exclusion Criteria:

* Known allergy to local anesthetics
* Known history of chronic pain disorders and/or chronic opioid use defined as > 10 mg of oral (PO) morphine or equivalent used daily for at least 30 days prior to enrollment
* Patient is a prisoner or incarcerated
* Significant liver disease that would inhibit prescription of opioids
* Significant kidney disease that would inhibit administration of gabapentin
* Patient has a history of opioid dependence requiring rehabilitation or the use of opioid antagonists
* Patient is pregnant
* Patients with a planned exploration with biopsies (no organs removed) will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Barroilhet, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Epidural Placement, ERP): Patients undergo epidural placement in the First Day Surgery pre-operative area or similar areas suitable for insertion of epidural catheters. In the post-operative anesthesia care unit, patients may receive medication via the epidural on an as needed basis, as determined by the anesthesia team. Dosing and rate of standardized medication will be managed by the anesthesia team until the epidural is removed. Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.
  Epidural analgesia: Receive epidural placement. Standard epidural medications and dosage are as follows:
  * 0.1% ropivicaine + 10 mcg/mL hydromorphone at 6 mL/hr continuous rate
  * 3 mL/hr RN bolus, to be used as needed based on pain ratings
  * 3 mL/30 minutes patient bolus, which is available on patient demand.
  Intraoperative Complication Management and Prevention: Undergo ERP
  Pain Therapy: Undergo ERP
Period: Overall Study
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Started | 52 | 52
Completed | 52 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP) | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 2 | 1 | 3
  30-39 years | 1 | 1 | 2
  40-49 years | 8 | 11 | 19
  50-59 years | 19 | 16 | 35
  60-69 years | 16 | 18 | 34
  70-79 years | 5 | 3 | 8
  80-89 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 51 | 49 | 100
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 48 | 48 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Relative Pain Scores, as Measured by the Pain Numeric Rating Scale (NRS)
Description: Relative pain scores between the epidural and non-epidural group will be analyzed by calculating a two-sided 95% confidence interval on the difference in mean scores between the two groups and concluding non-inferiority if this lies entirely below 2 points (mean non-epidural pain score proven, within a 95% confidence limit, to be at most 2 points worse than mean pain score in the epidural group). NRS rates pain on a 1-10 scale, with 1 being no pain, and 10 being the worst pain imaginable.
Time Frame: Up to 24 hours post-surgery
Population: Modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
score on a scale | 3.87 [3.35 to 4.38] | 4.95 [4.25 to 5.65]

2. Secondary Outcome: Average Daily Pain Score as Measured by Pain NRS Scores
Description: Will be compared using two-sided 95% confidence intervals for their mean differences. Superiority tests at the two-sided .05 level will be conducted by determining whether these confidence intervals overlap.
Time Frame: Up to 2 days following surgery
Population: modified intent to treat
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
score on a scale | 3.98 [3.27 to 4.42] | 5.12 [4.33 to 5.61]

3. Secondary Outcome: Difference in IL-2 Levels Between Pre-operative and Post-operative Values
Description: as for outcome 2
Time Frame: Baseline to up to day 1 post-surgery
Population: Modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 41 | 42
nmol/L | 9.6 [8.1 to 10.4] | 15.5 [14.0 to 16.3]

4. Secondary Outcome: Epidural Discontinuation Rates Prior to Planned Removal (in Epidural Group Only)
Description: Will be tabulated and presented for each group (where applicable).
Time Frame: Up to post-operative day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Epidural Placement, ERP)
Number analyzed (Participants) | 48
Participants | 4

5. Secondary Outcome: Length of Hospital Stay (Hours)
Description: as for outcome 2
Time Frame: From admission to time of discharge order placement
Population: Modified intent to treat
Measure: Mean (95% Confidence Interval); unit: hours
Groups:
- Enhanced Recovery Pathway: Patients complete the ERP comprising increased activity, dietary restrictions, fluid balance, as well as anti-nausea, anti-inflammatory and pain medications at specific times. Patients will have access to additional pain medications as needed to control their pain.
  Intraoperative Complication Management and Prevention: Undergo ERP
  Pain Therapy: Undergo ERP
Arm/Group | Arm I (Epidural Placement, ERP) | Enhanced Recovery Pathway
Number analyzed (Participants) | 52 | 45
hours | 99.83 [79.22 to 120.43] | 87.25 [73.45 to 101.05]

6. Secondary Outcome: Length of Time Until Return of Bowel Function
Description: as for outcome 2
Time Frame: From completion of surgery to passage of flatus (report in days)
Population: modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm I (Epidural Placement, ERP) | Enhanced Recovery Pathway
Number analyzed (Participants) | 51 | 46
days | 2.22 [1.91 to 2.52] | 2.20 [1.95 to 2.44]

7. Secondary Outcome: Number of Recorded Episodes of Emesis
Description: as for outcome 2
Time Frame: Up to 5 days post-surgery
Population: modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
number of episodes | .192 [.046 to .339] | .1875 [.045 to .330]

8. Secondary Outcome: Patient Satisfaction Scores Related to Pain Metrics, as Measured by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey
Description: Will be compared using two-sided 95% confidence intervals for their mean differences. Superiority tests at the two-sided .05 level will be conducted by determining whether these confidence intervals overlap. Scores range from 1 to 4, with higher scores indicating higher satisfaction.
Time Frame: At 4 weeks post-operative visit
Population: Modified intent to treat
Measure: Mean (95% Confidence Interval); unit: score on a scale of 1-4
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 46 | 39
score on a scale of 1-4 | 3.78 [3.65 to 3.90] | 3.87 [3.76 to 3.98]

9. Secondary Outcome: Post-operative Antiemetic Use (Measured in mg of Ondanestron Used in the First 24 Hours After Surgery)
Description: as for outcome 2
Time Frame: Up to 4 weeks post-surgery
Population: modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
mg | 4.46 [3.02 to 5.90] | 3.17 [2.04 to 4.29]

10. Secondary Outcome: Post-operative Complications (UTIs, Thromboembolic Events, Pneumonia, Blood Transfusion, Myocardial Infarction, Falls)
Description: # of events in each group will be reported
Time Frame: Up to 6 weeks post-surgery
Population: modified intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
Participants | 15 | 12

11. Secondary Outcome: Readmission Rate
Description: as for outcome 2
Time Frame: Up to 6 weeks post-surgery
Population: modified intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
Participants | 2 | 2

12. Secondary Outcome: Total Opioid Use Measured in Oral Morphine Equivalents (mg)
Description: as for outcome 2
Time Frame: Up to first 2 days post-surgery
Population: Modified intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
Number analyzed (Participants) | 52 | 48
mg | 50.1 [34.48 to 65.72] | 82.56 [63.13 to 101.97]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Arm I (Epidural Placement, ERP) | Arm II (ERP)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/52
Other Adverse Events (participants affected / at risk) | 35/52 | 28/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Epidural Placement, ERP) (N=52) | Arm II (ERP) (N=52)
wound infection, fascial dehiscence (Infections and infestations) | 1 (1) | 0 (0) — required second surgery
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — requiring IV antibiotics and hospital readmission
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Epidural Placement, ERP) (N=52) | Arm II (ERP) (N=52)
anemia (Blood and lymphatic system disorders) | 35 (35) | 28 (28)
vascular thrombolic event (Blood and lymphatic system disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Cytokine samples were not able to be interpreted due to huge variances, and they are being run again on a different flow cytometry machine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02423876/Prot_SAP_000.pdf